CLINICAL TRIAL: NCT03951805
Title: A Trial Comparing NNC0148-0287 C (Insulin 287) Versus Insulin Glargine U100, Both in Combination With Metformin, With or Without DPP4 Inhibitors and With or Without SGLT2 Inhibitors, in Insulin-naïve Subjects With Type 2 Diabetes Mellitus
Brief Title: A Research Study to Compare Two Types of Insulin: Insulin 287 and Insulin Glargine in People With Type 2 Diabetes Who Have Not Used Insulin Before
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1436-4465; U1111-1219-5474 (Other: World Health Organization (WHO)); 2018-003406-11 (EudraCT Number)
Record Dates: First submitted 2019-05-10; First posted 2019-05-15 (Actual); Results first posted 2021-01-08 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin icodec; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Insulin 287 algorithm A (Experimental): Controlled on metformin with or without DPP4i (dipeptidyl peptidase-4 inhibitors) and with or without SGLT2i (sodium-glucose cotransporter 2 inhibitors).
  Interventions: Drug: Insulin icodec
- Insulin 287 algorithm B (Experimental): Controlled on metformin with or without DPP4i and with or without SGLT2i.
  Interventions: Drug: Insulin icodec
- Insulin 287 algorithm C (Experimental): Controlled on metformin with or without DPP4i and with or without SGLT2i.
  Interventions: Drug: Insulin icodec
- Insulin Glargine algorithm D (Active Comparator): Controlled on metformin with or without DPP4i and with or without SGLT2i.
  Interventions: Drug: Insulin Glargine

INTERVENTIONS:
Drug: Insulin icodec — Administered subcutaneously SC once weekly. Starting dose will be 70U.
  Other Names: Insulin 287
  Arms: Insulin 287 algorithm A; Insulin 287 algorithm B; Insulin 287 algorithm C
Drug: Insulin Glargine — Administered subcutaneously SC once daily.The starting dose will be 10U.
  Arms: Insulin Glargine algorithm D

SUMMARY:
This study compares insulin 287 (a possible new medicine) to insulin glargine (a medicine doctors can already prescribe) in people with type 2 diabetes. Different ways of changing the dose of insulin 287 are also compared. This is done to find the best way to change the dose of insulin 287. Participants will either get insulin 287 that they will have to inject once a week or insulin glargine that participants will have to inject once a day. Which treatment participants get is decided by chance. The study will last for about 5 months (23 weeks). Participants will have 14 clinic visits and 6 phone calls with the study doctor. At 3 of the clinic visits participants will be asked not to eat or drink anything (except for water) in the last 8 hours before the visit. During the study, the study doctor will ask participants to:

* measure blood sugar every day with a blood sugar meter using a finger prick.
* write down different information in a diary daily and return this to the study doctor.
* wear a medical device (sensor) that measure blood sugar all the time for 18 weeks (about 4 months) during the study.

Women cannot take part if pregnant, breastfeeding or plan to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-75 years (both inclusive) at the time of signing informed consent
* Diagnosed with type 2 diabetes mellitus greater than or equal to 180 days prior to the day of screening
* HbA1c of 7.0-10.0% (53.0-85.8 mmol/mol) (both inclusive) as assessed by central laboratory
* Stable daily dose(s) for 90 days prior to the day of screening of any of the following antidiabetic drug(s) or combination regime(s):

  1. Any metformin formulations greater than or equal to 1500 mg or maximum tolerated or effective dose (as documented in subject's medical records)
  2. Free or fixed combination therapy: Metformin as outlined above plus/minus DPP4i with or without SGLT2i is allowed:

  i) DPP4i (greater than or equal to half of the maximum approved dose according to local label or maximum tolerated or effective dose) ii) SGLT2i (greater than or equal to half of the maximum approved dose according to local label or maximum tolerated or effective dose )
* Insulin-naïve. However, short term insulin treatment for a maximum of 14 days prior to the day of screening is allowed, as is prior insulin treatment for gestational diabetes
* Body mass index (BMI) below or equal to 40.0 kg/m^2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2020-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (42):
- United States (11):
  - Novo Nordisk Investigational Site, Anaheim, California
  - Novo Nordisk Investigational Site, Lancaster, California
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Statesboro, Georgia
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, West Seneca, New York
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Austin, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Schertz, Texas
- Croatia (4):
  - Novo Nordisk Investigational Site, Karlovac
  - Novo Nordisk Investigational Site, Osijek
  - Novo Nordisk Investigational Site, Rijeka
  - Novo Nordisk Investigational Site, Varaždin
- Germany (9):
  - Novo Nordisk Investigational Site, Bad Mergentheim
  - Novo Nordisk Investigational Site, Essen
  - Novo Nordisk Investigational Site, Falkensee
  - Novo Nordisk Investigational Site, Friedrichsthal
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Münster
  - Novo Nordisk Investigational Site, Oldenburg I. Holst
  - Novo Nordisk Investigational Site, Pohlheim
  - Novo Nordisk Investigational Site, Saint Ingbert-Oberwürzbach
- Hungary (3):
  - Novo Nordisk Investigational Site, Kaposvár
  - Novo Nordisk Investigational Site, Szeged
  - Novo Nordisk Investigational Site, Zalaegerszeg
- Poland (5):
  - Novo Nordisk Investigational Site, Bialystok
  - Novo Nordisk Investigational Site, Lublin
  - Novo Nordisk Investigational Site, Radom
  - Novo Nordisk Investigational Site, Tomaszów Mazowiecki
  - Novo Nordisk Investigational Site, Warsaw
- Slovakia (6):
  - Novo Nordisk Investigational Site, Banská Bystrica
  - Novo Nordisk Investigational Site, Košice
  - Novo Nordisk Investigational Site, Nitra
  - Novo Nordisk Investigational Site, Rimavská Sobota
  - Novo Nordisk Investigational Site, Rožňava
  - Novo Nordisk Investigational Site, Veľký Meder
- Spain (4):
  - Novo Nordisk Investigational Site, A Coruña
  - Novo Nordisk Investigational Site, Barakaldo
  - Novo Nordisk Investigational Site, La Roca Del Vallés
  - Novo Nordisk Investigational Site, Vic (Barcelona)

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Lingvay I, Buse JB, Franek E, Hansen MV, Koefoed MM, Mathieu C, Pettus J, Stachlewska K, Rosenstock J. A Randomized, Open-Label Comparison of Once-Weekly Insulin Icodec Titration Strategies Versus Once-Daily Insulin Glargine U100. Diabetes Care. 2021 Jul;44(7):1595-1603. doi: 10.2337/dc20-2878. Epub 2021 Apr 19. PMID 33875484

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 38 sites in 7 countries as follows: Croatia (4), Germany (9), Hungary (3), Poland (4), Slovakia (5), Spain (4), United States (9). In addition, 1 site in Slovakia and 3 sites in the United States screened, but didn't randomise any subjects.
Pre-assignment Details: Participants were randomised to receive once weekly insulin 287 using one of 3 different titration algorithms (A, B, C), or once daily insulin glargine (titration algorithm D); as add-on to background therapy with metformin with or without dipeptidyl peptidase-4 inhibitors (DPP4i) and with or without sodium-glucose cotransporter 2 inhibitors (SGLT2i).
Groups:
- Insulin 287 (Titration Algorithm A): Participants were to receive once weekly subcutaneous (s.c.) injection of insulin 287 for 16 weeks, using PDS290 prefilled pen-injector at a starting dose of 70 units (U). The dose was adjusted weekly during the treatment period using titration algorithm A with American Diabetes Association (ADA) glycaemic target of 4.4-7.2 mmol/L (80-130 mg/dL), based on 3 pre-breakfast self-measured plasma glucose (SMPG) values measured on 2 previous days and on the day of the contact. If at least one pre-breakfast SMPG value was: < 4.4 mmol/L: insulin dose reduced by 21 U. Otherwise, the dose adjustment was based on the mean of SMPG values. If the mean was between 4.4-7.2 mmol/L: no adjustment; > 7.2 mmol/L: insulin dose increased by 21 U. All participants used metformin with or without DPP4i and with or without SGLT2i at the stable, pre-trial dose and at the same frequency during the entire treatment period unless due to safety concerns related to the background medication.
- Insulin 287 (Titration Algorithm B): Participants were to receive once weekly s.c. injection of insulin 287 for 16 weeks, using PDS290 prefilled pen-injector at a starting dose of 70 U. The dose was adjusted weekly during the treatment period using titration algorithm B with ADA glycaemic target of 4.4-7.2 mmol/L (80-130 mg/dL), based on 3 pre-breakfast SMPG values measured on 2 previous days and on the day of the contact. If at least one pre-breakfast SMPG value was: < 4.4 mmol/L: insulin dose reduced by 28 U. Otherwise, the dose adjustment was based on the mean of SMPG values. If the mean was between 4.4-7.2 mmol/L: no adjustment; > 7.2 mmol/L: insulin dose increased by 28 U. All participants used metformin with or without DPP4i and with or without SGLT2i at the stable, pre-trial dose and at the same frequency during the entire treatment period unless due to safety concerns related to the background medication
- Insulin 287 (Titration Algorithm C): Participants were to receive once weekly s.c. injection of insulin 287 for 16 weeks, using PDS290 prefilled pen-injector at a starting dose of 70 U. The dose was adjusted weekly during the treatment period using titration algorithm C with glycaemic target of 3.9-6.0 mmol/L (70-108 mg/dL), based on 3 pre-breakfast SMPG values measured on 2 previous days and on the day of the contact. If at least one pre-breakfast SMPG value was: < 3.9 mmol/L: insulin dose reduced by 28 U. Otherwise, the dose adjustment was based on the mean of SMPG values. If the mean was between 3.9-6.0 mmol/L: no adjustment; > 6.0 mmol/L: insulin dose increased by 28 U. All participants used metformin with or without DPP4i and with or without SGLT2i at the stable, pre-trial dose and at the same frequency during the entire treatment period unless due to safety concerns related to the background medication.
- Insulin Glargine (Titration Algorithm D): Subjects were to receive once daily s.c. injection of Insulin glargine for 16 weeks, using SoloSTAR pre-filled pen-injector at a starting dose of 10 U. The dose was adjusted weekly during the treatment period using titration algorithm D with ADA glycaemic target of 4.4-7.2 mmol/L (80-130 mg/dL), based on 3 pre-breakfast SMPG values measured on 2 previous days and on the day of the contact. If at least one pre-breakfast SMPG value was: < 4.4 mmol/L: insulin dose reduced by 4 U. Otherwise, the dose adjustment was based on the mean of SMPG values. If the mean was between 4.4-7.2 mmol/L: no adjustment; > 7.2 mmol/L: insulin dose increased by 4 U. All subjects used metformin with or without DPP4i and with or without SGLT2i at the stable, pre-trial dose and at the same frequency during the entire treatment period unless due to safety concerns related to the background medication.
Period: Overall Study
Arm/Group | Insulin 287 (Titration Algorithm A) | Insulin 287 (Titration Algorithm B) | Insulin 287 (Titration Algorithm C) | Insulin Glargine (Titration Algorithm D)
Started | 51 | 51 | 52 | 51
Full Analysis Set (FAS) | 51 | 51 | 52 | 51
Safety Analysis Set (SAS) | 51 | 51 | 52 | 51
Completed | 50 | 51 | 52 | 51
Not Completed | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set included all randomised participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin 287 (Titration Algorithm A) | Insulin 287 (Titration Algorithm B) | Insulin 287 (Titration Algorithm C) | Insulin Glargine (Titration Algorithm D) | Total
Number analyzed (Participants) | 51 | 51 | 52 | 51 | 205
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (9.1) | 61.2 (8.0) | 61.4 (8.0) | 60.2 (8.1) | 60.7 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 23 | 24 | 24 | 95
  Male | 27 | 28 | 28 | 27 | 110
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 2 | 3 | 12
  Not Hispanic or Latino | 49 | 46 | 50 | 48 | 193
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 2 | 0 | 0 | 2
  Black or African American | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 1 | 1
  White | 51 | 49 | 51 | 47 | 198
  other | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time in Target Range (TIR) 3.9-10.0 Millimoles Per Liter (mmol/L) (70-180 Milligrams Per Deciliter (mg/dL) Measured Using CGM (Continuous Glucose Monitoring)
Description: The percentage of time spent in glycaemic target range was calculated as 100 times the number of recorded measurements in glycaemic target range 3.9-10.0 mmol/L (70-180 mg/dL), both inclusive divided by the total number of recorded measurements. The endpoint was evaluated based on the data from the on-treatment without rescue medication observation period, which was the time period when a participant was considered exposed to trial product, excluding any period after initiation of a non-randomised insulin treatment (rescue medication). The endpoint is based on data recorded by CGM system. It was required that at least 70% of the planned CGM measurements during weeks 15-16 were available for endpoint data to be included in the analysis.
Time Frame: During the last 2 weeks of treatment (week 15 and 16)
Population: Full analysis set included all randomised participants. Overall number of participants analyzed = Number of participants who contributed to the analysis.
Measure: Least Squares Mean (Standard Error); unit: Percentage of time
Arm/Group | Insulin 287 (Titration Algorithm A) | Insulin 287 (Titration Algorithm B) | Insulin 287 (Titration Algorithm C) | Insulin Glargine (Titration Algorithm D)
Number analyzed (Participants) | 51 | 51 | 51 | 50
Percentage of time | 76.65 (1.81) | 82.97 (1.80) | 80.89 (1.81) | 75.89 (1.82)
Statistical Analysis 1: Comparison: Insulin 287 (Titration Algorithm A) vs Insulin Glargine (Titration Algorithm D); The response and change from baseline in response during the last two weeks of treatment (week 15 and 16) are analysed using an analysis of covariance (ANCOVA) model with treatment and SGLT2i use as fixed factors, and baseline response as covariate. Missing endpoint values are imputed using multiple imputation based on own treatment arm with baseline response as a covariate. Each imputed dataset is analysed separately and estimates are combined using Rubin's rules; Test type: Other; p = 0.7675, ANCOVA; Treatment difference = 0.76, 95% CI 2-sided [-4.28 to 5.80]
Statistical Analysis 2: Comparison: Insulin 287 (Titration Algorithm B) vs Insulin Glargine (Titration Algorithm D); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0051, ANCOVA; Treatment difference = 7.08, 95% CI 2-sided [2.12 to 12.04]
Statistical Analysis 3: Comparison: Insulin 287 (Titration Algorithm C) vs Insulin Glargine (Titration Algorithm D); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0519, ANCOVA; Treatment difference = 5.01, 95% CI 2-sided [-0.04 to 10.05]

2. Secondary Outcome: Change in HbA1c (Glycated Haemoglobin)
Description: Estimated mean change in HbA1c from baseline (week 0, visit 2) to end of treatment (week 16, visit 18) is presented. The endpoint was evaluated based on the data from the on-treatment without rescue medication observation period, which was the time period when a participant was considered exposed to trial product, excluding any period after initiation of a non-randomised insulin treatment (rescue medication).
Time Frame: From baseline week 0 (visit 2) to week 16 (visit 18)
Population: Full analysis set included all randomised participants.
Measure: Least Squares Mean (Standard Error); unit: Percentage point of HbA1c
Arm/Group | Insulin 287 (Titration Algorithm A) | Insulin 287 (Titration Algorithm B) | Insulin 287 (Titration Algorithm C) | Insulin Glargine (Titration Algorithm D)
Number analyzed (Participants) | 51 | 51 | 52 | 51
Percentage point of HbA1c | -1.00 (0.08) | -1.22 (0.08) | -1.38 (0.08) | -1.02 (0.08)

3. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Estimated mean change in FPG from baseline (week 0, visit 2) to end of treatment (week 16, visit 18) is presented. The endpoint was evaluated based on the data from the on-treatment without rescue medication observation period, which was the time period when a participant was considered exposed to trial product, excluding any period after initiation of a non-randomised insulin treatment (rescue medication).
Time Frame: From baseline week 0 (visit 2) to week 16 (visit 18)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Millimoles per liter (mmol/L)
Arm/Group | Insulin 287 (Titration Algorithm A) | Insulin 287 (Titration Algorithm B) | Insulin 287 (Titration Algorithm C) | Insulin Glargine (Titration Algorithm D)
Number analyzed (Participants) | 51 | 50 | 51 | 49
Millimoles per liter (mmol/L) | -2.23 (0.17) | -2.42 (0.17) | -3.01 (0.17) | -2.34 (0.17)

4. Secondary Outcome: Change in Body Weight
Description: Estimated mean change in body weight from baseline (week 0, visit 2) to end of treatment (week 16, visit 18) is presented. The endpoint was evaluated based on the data from the on-treatment without rescue medication observation period, which was the time period when a participant was considered exposed to trial product, excluding any period after initiation of a non-randomised insulin treatment (rescue medication).
Time Frame: From baseline week 0 (visit 2) to week 16 (visit 18)
Population: Full analysis set included all randomised participants.
Measure: Least Squares Mean (Standard Error); unit: Kilogram (Kg)
Arm/Group | Insulin 287 (Titration Algorithm A) | Insulin 287 (Titration Algorithm B) | Insulin 287 (Titration Algorithm C) | Insulin Glargine (Titration Algorithm D)
Number analyzed (Participants) | 51 | 51 | 52 | 51
Kilogram (Kg) | 0.87 (0.35) | 1.11 (0.35) | 1.25 (0.35) | 0.63 (0.35)

5. Secondary Outcome: Weekly Insulin Dose
Description: Estimated mean average weekly insulin dose during the last 2 weeks of treatment is presented. The endpoint was evaluated based on the data from the on-treatment without rescue medication observation period, which was the time period when a participant was considered exposed to trial product, excluding any period after initiation of a non-randomised insulin treatment (rescue medication).
Time Frame: During the last 2 weeks of treatment (week 15 and 16)
Population: Full analysis set included all randomised participants.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units of insulin (U)
Arm/Group | Insulin 287 (Titration Algorithm A) | Insulin 287 (Titration Algorithm B) | Insulin 287 (Titration Algorithm C) | Insulin Glargine (Titration Algorithm D)
Number analyzed (Participants) | 51 | 51 | 52 | 51
Units of insulin (U) | 142.47 [119.78 to 169.45] | 176.38 [148.30 to 209.78] | 208.90 [175.94 to 248.04] | 145.56 [122.38 to 173.12]

6. Secondary Outcome: Number of Treatment Emergent Adverse Events (TEAEs)
Description: A TEAE was defined as an event that had onset date (or increase in severity) during the on-treatment observation period. The on-treatment observation period was the time period from first dose of trial product (week 0, visit 2) until the follow-up visit (week 21, visit 20) or the last date on trial product + 5 weeks for once daily insulin and +6 weeks for once weekly insulin.
Time Frame: From baseline week 0 (visit 2) to week 21 (visit 20)
Population: Safety analysis set included all participants exposed to at least one dose of trial product.
Measure: Number; unit: Count of events
Arm/Group | Insulin 287 (Titration Algorithm A) | Insulin 287 (Titration Algorithm B) | Insulin 287 (Titration Algorithm C) | Insulin Glargine (Titration Algorithm D)
Number analyzed (Participants) | 51 | 51 | 52 | 51
Count of events | 44 | 67 | 58 | 45

7. Secondary Outcome: Number of Severe Hypoglycaemic Episodes (Level 3)
Description: Severe hypoglycaemic episodes (level 3) were defined as episodes that were associated with severe cognitive impairment requiring external assistance for recovery. Number of severe hypoglycaemic episodes that occurred from baseline (week 0, visit 2) to end of treatment (week 16, visit 18) are presented.
Time Frame: From baseline week 0 (visit 2) to week 16 (visit 18)
Population: Safety analysis set included all participants exposed to at least one dose of trial product.
Measure: Number; unit: Count of events
Arm/Group | Insulin 287 (Titration Algorithm A) | Insulin 287 (Titration Algorithm B) | Insulin 287 (Titration Algorithm C) | Insulin Glargine (Titration Algorithm D)
Number analyzed (Participants) | 51 | 51 | 52 | 51
Count of events | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Clinically Significant Hypoglycaemic Episodes (Level 2) (Below 3.0 mmol/L (54 Milligrams Per Deciliter [mg/dL]), Confirmed by Blood Glucose (BG) Meter) or Severe Hypoglycaemic Episodes (Level 3)
Description: Clinically significant hypoglycaemic episodes (level 2) were defined as episodes that were sufficiently low to indicate serious, clinically important hypoglycaemia with plasma glucose value of less than (<) 3.0 mmol/L (54 mg/dL). Severe hypoglycaemic episodes (level 3) were defined as episodes that were associated with severe cognitive impairment requiring external assistance for recovery. Number of clinically significant hypoglycaemic episodes (level 2), confirmed by blood glucose (BG) meter or severe hypoglycaemic episodes (level 3) that occured from baseline (week 0, visit 2) to end of treatment (week 16, visit 18) are presented.
Time Frame: From baseline week 0 (visit 2) to week 16 (visit 18)
Population: Safety analysis set included all participants exposed to at least one dose of trial product.
Measure: Number; unit: Count of events
Arm/Group | Insulin 287 (Titration Algorithm A) | Insulin 287 (Titration Algorithm B) | Insulin 287 (Titration Algorithm C) | Insulin Glargine (Titration Algorithm D)
Number analyzed (Participants) | 51 | 51 | 52 | 51
Count of events | 1 | 2 | 8 | 0

9. Secondary Outcome: Number of Hypoglycaemic Alert Episodes (Level 1) (Greater Than or Equal to 3.0 and Below 3.9 mmol/L (Greater Than or Equal to 54 and Below 70 mg/dL), Confirmed by Blood Glucose (BG) Meter)
Description: Hypoglycaemia alert value (level 1) was defined as episodes that were sufficiently low for treatment with fast-acting carbohydrate and dose adjustment of glucose-lowering therapy with plasma glucose value of equal to or above (>=) 3.0 and < 3.9 mmol/L (>= 54 and < 70 mg/dL) confirmed by BG meter. Number of hypoglycaemic alert episodes (level 1) that occured from baseline (week 0, visit 2) to end of treatment (week 16, visit 18) are presented.
Time Frame: From baseline week 0 (visit 2) to week 16 (visit 18)
Population: Safety analysis set included all participants exposed to at least one dose of trial product.
Measure: Number; unit: Count of events
Arm/Group | Insulin 287 (Titration Algorithm A) | Insulin 287 (Titration Algorithm B) | Insulin 287 (Titration Algorithm C) | Insulin Glargine (Titration Algorithm D)
Number analyzed (Participants) | 51 | 51 | 52 | 51
Count of events | 14 | 20 | 110 | 10

ADVERSE EVENTS:
Time Frame: From baseline (week 0) to week 21 Results are based on the safety analysis set which included all participants exposed to at least one dose of trial product.
Description: All presented adverse events are treatment emergent adverse events (TEAEs). TEAE was defined as an event that had onset date (or increase in severity) during the on-treatment observation period. The on-treatment observation period was the time period from first dose of trial product until the follow-up visit or the last date on trial product + 5 weeks for once daily insulin and +6 weeks for once weekly insulin.
Arm/Group | Insulin 287 (Titration Algorithm A) | Insulin 287 (Titration Algorithm B) | Insulin 287 (Titration Algorithm C) | Insulin Glargine (Titration Algorithm D)
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51 | 0/52 | 0/51
Serious Adverse Events (participants affected / at risk) | 3/51 | 1/51 | 0/52 | 2/51
Other Adverse Events (participants affected / at risk) | 9/51 | 10/51 | 7/52 | 9/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin 287 (Titration Algorithm A) (N=51) | Insulin 287 (Titration Algorithm B) (N=51) | Insulin 287 (Titration Algorithm C) (N=52) | Insulin Glargine (Titration Algorithm D) (N=51)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Choroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin 287 (Titration Algorithm A) (N=51) | Insulin 287 (Titration Algorithm B) (N=51) | Insulin 287 (Titration Algorithm C) (N=52) | Insulin Glargine (Titration Algorithm D) (N=51)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (3) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 5 (7) | 2 (3)
Nasopharyngitis (Infections and infestations) | 5 (7) | 7 (7) | 2 (2) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/05/NCT03951805/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/05/NCT03951805/SAP_001.pdf